CLINICAL TRIAL: NCT04931290
Title: Supracapsular Ahmed Glaucoma Valve Plate Delivery Technique for Management of Encapsulated Bleb in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Dina abdelfattah, Lecturer of ophthalmology, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.21.03.1246.R1.R2
Record Dates: First submitted 2021-06-12; First posted 2021-06-18 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- supracapsular delivery of plate of valve (Experimental): ncision of the perilimbal superior temporal conjunctiva with separation of the conjunctiva from the Tenon's capsule till reaching the encapsulated valve plate. Incision of the capsule in a z pattern will be done then the plate is dissected from the tissues and delivered out of the capsule through the opening to the subconjunctival space.The mobility of AGV and its tube will be evaluated and refixation of the plate will be done if needed. The plate will be covered with ologen implant sizing 12mm width and 1 mm thickness. The conjunctiva will be closed by 10/0 nylon sutures.
  Interventions: Procedure: Supracapsular Ahmed Glaucoma Valve plate delivery technique

INTERVENTIONS:
Procedure: Supracapsular Ahmed Glaucoma Valve plate delivery technique — incision of the perilimbal superior temporal conjunctiva with separation of the conjunctiva from the Tenon's capsule till reaching the encapsulated valve plate. Incision of the capsule in a z pattern will be done then the plate is dissected from the tissues and delivered out of the capsule through the opening to the subconjunctival space.The mobility of AGV and its tube will be evaluated and refixation of the plate will be done if needed. The plate will be covered with ologen implant sizing 12mm width and 1 mm thickness. The conjunctiva will be closed by 10/0 nylon sutures.

SUMMARY:
This study aims to assess the safety and efficacy of supracapsular Ahmed Glaucoma Valve plate delivery for management of encapsulated bleb in pediatric patients with failed Ahmed Glaucoma Valve.

This is a prospective interventional study. It will be conducted in Mansoura University in the duration from April 2020 to January 2021. The study will include pediatric patients less than 18 years with failed AGV with encapsulated bleb and high IOP above 21 mm Hg in two consecutive visits inspite of topical glaucoma medications

DETAILED DESCRIPTION:
Introduction Refractory glaucoma is a complicated type of glaucoma that is characterized by high intraocular pressure (IOP), making it difficult to treat by traditional medical or surgical therapies. Trabeculectomy has shown poor long-term outcomes for refractory glaucoma, making shunt surgery a better alternative. [1]Ahmed glaucoma valve (AGV) is effective procedure in management of refractory glaucoma with long-term follow-up in Egyptian patients.[2] AGV, a shunt device, is used either initially or after conventional procedures fail to treat refractory glaucoma. It helps the aqueous humor flow directly into the silicone tube.[3] Encapsulation of the AGV is an early complication especially in pediatric patients leading to postoperative elevation of intraocular pressure [4]. Encapsulation inhibits the fluid drainage leading to failure of the procedure. The valve mechanism is blocked by contracted scar tissue, but the device itself is not affected by the encapsulation..[5] The reasons for this excessive fibrotic reaction and capsule impermeability are not fully understood. Apart from implant properties, such as size, shape, surface properties and biomaterial other mechanisms leading to collagen distribution, proliferation and adhesion of fibroblasts have been suggested to contribute to the encapsulation process .[6]

Different techniques were developed for revision of this encapsulated bleb. Surgical excision of the capsule immediately leads to an aqueous flow and drop of intraocular pressure [4, 7], but it carries the risk of reformation of the capsule again. Bleb needle revision is another method that targets the fibrosis tissue and has long been employed in the treatment of encapsulated bleb following trabeculectomy. Despite the favorable outcomes after trabeculectomy, this modality is not generally used after AGV implantation. A few reports have investigated the application of needle revision in AGVs[8] Using antimetabolites as mitomycin c and 5-FU during needling over the plate of an AGV may also be an effective and safe choice in patients with elevated IOP due to encapsulation or fibrosis.[9] Aim of the Study This study aims to assess the safety and efficacy of supracapsular Ahmed Glaucoma Valve plate delivery for management of encapsulated bleb in pediatric patients with failed Ahmed Glaucoma Valve.

Patient and methods This is a prospective interventional study. It will be conducted in Mansoura University in the duration from April 2020 to January 2021. The study will include pediatric patients less than 18 years with failed AGV with encapsulated bleb and high IOP above 21 mm Hg in two consecutive visits inspite of topical glaucoma medications. Patients with intraocular inflammations or ocular surface diseases will be excluded from the study.

The outcome will be measured as IOP and its association with the number of postoperative glaucoma medications. IOP ≤ 21 mmHg without medications indicates complete success while IOP ≤ 21 mmHg with medications indicates qualified success, an IOP <6 mmHg i defined as hypotony and IOP above 21 mm Hg with medications indicates failure Cooperative patients will preoperatively be subjected to IOP measurement using hand held Perkin's applanation tonometer, visual acuity (VA) assessment using a Snellen E chart, optic disc examination by a Volk+90 lens, slit lamp examination for assessment of corneal clarity, and assessment for any corneal tube-touch and measurement of anterior chamber depth. Examination under anesthesia will be done in younger or uncooperative children.

The following operative technique will be followed: incision of the perilimbal superior temporal conjunctiva with separation of the conjunctiva from the Tenon's capsule till reaching the encapsulated valve plate. Incision of the capsule in a z pattern will be done then the plate is dissected from the tissues and delivered out of the capsule through the opening to the subconjunctival space.The mobility of AGV and its tube will be evaluated and refixation of the plate will be done if needed. The plate will be covered with ologen implant sizing 12mm width and 1 mm thickness. The conjunctiva will be closed by 10/0 nylon sutures.

A postoperative treatment course of combined antibiotic and steroid eye drops every four hours in the first week, gradually tapered over the next 2 weeks, will be prescribed. IOP, VA, and optic disc examination by Volk+90 lens, and slit lamp examination will be performed at the follow-up period at 1st day, 1st week , 1st month and 3rd month postoperatively.

Ethical Consideration:

Study protocol is approved by medical research ethics committee, faculty of medicine, Mansoura University.Informed written consent will be obtained from each patient's parents after being informed of the risks, benefits, and alternatives of surgery. The confidentiality of participant data is ensured. The participants are free not to participate or to leave the research at any time, without penalty Statistical analysis Statistical analyses will be carried out using the Statistical Package for Social Sciences (SPSS 19.0 for windows, SPSS Inc, Chicago, IL, USA). Results will be considered statistically significant when P is < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients less than 18 years with failed AGV with encapsulated bleb and high IOP above 21 mm Hg in two consecutive visits inspite of topical glaucoma medications

Exclusion Criteria:

* intraocular inflammations or ocular surface diseases

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 6 month
  IOP
success rates | 6 month
  IOP ≤ 21 mmHg without medications indicates complete success while IOP ≤ 21 mmHg with medications indicates qualified success, an IOP <6 mmHg i defined as hypotony and IOP above 21 mm Hg with medications indicates failure

CONTACTS AND LOCATIONS:
Overall Officials: Dina AbdElfattah, MD, Principal Investigator — Mansoura University
Locations (1):
- Dina Abd Elfattah, Al Mansurah, Dakahlia Governorate, Egypt